CLINICAL TRIAL: NCT05812911
Title: An Adaptive Randomized Controlled Trial (RCT) Comparing High-flow Nasal Cannula Oxygen and Noninvasive Ventilation to Standard Oxygenation in Non-selected Intensive Care Unit Patients Admitted for Hypoxemic Acute Respiratory Failure: The KISS Trial (Key Oxygenation Interventions in Surgical and Non-Surgical Patients)
Brief Title: Comparing High-flow Nasal Cannula Oxygen and Noninvasive Ventilation to Standard Oxygenation in Non-selected ICU Patients Admitted for Hypoxemic ARF
Acronym: KISS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL20_0031
Record Dates: First submitted 2023-03-31; First posted 2023-04-14 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Acute Respiratory Failure
Keywords: High-Flow Nasal Cannula Oxygen; Non-Invasive Ventilation; Post-Operative; Immunocompromised; Acute Respiratory Failure; Intensive Care Unit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard oxygen therapy (Active Comparator): Patients will receive standard oxygen. First attempt device in usual care.
  Interventions: Procedure: Standard oxygen
- High-Flow nasal cannula therapy (HFNO) (Experimental): Patient will receive HFNO using a humidification system or via the high-flow interface of the ICU ventilator.
  Interventions: Procedure: HFNO
- Noninvasive ventilation therapy (NIV) (Experimental): Between NIV sessions, patients will receive HFNO with the same modalities than the HFNO group.
  Interventions: Procedure: NIV

INTERVENTIONS:
Procedure: Standard oxygen — Standard oxygen therapy administered through a Venturi mask allowing a fraction of inspired oxygen (FiO2) setting to maintain a peripheral oxygen saturation (SpO2) ≥ 94%.
  For medical reasons left to the clinician appreciation (such as a COPD or pulmonary fibrosis or other conditions), a SpO2 ≥ 90% will be accepted.
  Arms: Standard oxygen therapy
Procedure: HFNO — The oxygen therapy will be administered in a semi-sitting position, with a setting of the FiO2 and the oxygen flow rate, to obtain a SpO2 ≥ 94%.
  For medical reasons left to the clinician appreciation (such as a COPD or pulmonary fibrosis or other conditions), a SpO2 ≥ 90% will be accepted.
  Arms: High-Flow nasal cannula therapy (HFNO)
Procedure: NIV — Systematic application of NIV using two levels of pressure, pressure support (PS) + positive end-expiratory pressure (PEEP) provided using a dedicated NIV ventilator or a standard ICU ventilator with the " NIV module " through a facial mask. The FiO2 will be set to obtain a SpO2 ≥ 94%.
  For medical reasons left to the clinician appreciation (such as a COPD or pulmonary fibrosis or other conditions), a SpO2 ≥ 90% will be accepted.
  Arms: Noninvasive ventilation therapy (NIV)

SUMMARY:
The goal of this clinical trial is to determine whether one of the two oxygenation or ventilation strategies (NIV and/or HFNO) is superior to standard oxygen to reduce 28-day mortality rate in hypoxemic acute respiratory failure (ARF) patients.

DETAILED DESCRIPTION:
This randomized controlled trial is a superiority study to test if one of the methods (NIV and/or HFNO) is superior to standard oxygen in ARF patients requiring oxygen. It is an investigator-initiated, multicenter, adaptive, three arms parallel-group trial with a computer-generated allocation sequence and an electronic system-based randomization, with a stratification on medical (then stratification between immunocompromised and non-immunocompromised patients) versus surgical (then stratification between cardiothoracic and abdominal patients).

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years)
* A diagnosis of hypoxemic ARF occurring defined as the presence and persistence for more than 30 minutes of hypoxemia (defined by a partial oxygen pressure <60 mm Hg when breathing room air or <80 mmHg when breathing 15 L/min of oxygen or a peripheral oxygen saturation [SpO2] ≤90% when breathing room air and/or a PaO2(partial pressure of oxygen)/FiO2 ratio < 300 mmHg plus either [1] a respiratory rate higher than 30/min or [2] clinical signs suggestive of intense respiratory muscle work and/or labored breathing, such as use of accessory respiratory muscles, paradoxical motion of the abdomen, or intercostal retraction).

Exclusion Criteria:

* Contraindications to NIV and/or HFNO
* Sleep apnea syndrome with home ventilator
* Immediate tracheal intubation
* Requirement for an emergent surgical procedure requiring intubation
* Hypercapnia with a formal indication for NIV (formal indication for NIV with PaCO2 ≥ 50 mmHg or clinical signs of hypercapnia)
* Isolated cardiogenic pulmonary edema (formal indication for NIV). Patients with pulmonary edema associated with another ARF etiology can be included.
* Anatomical factors precluding the use of NIV and/or HFNO
* Patients with limitation or withdrawal of life-sustaining therapies with a do-not-intubate order
* Pregnancy in progress or planned during the study period or breastfeeding women
* Patients protected by law (Art. L1121-6 and L1121-8 of the Code de la Santé Publique): Adult protected by law or patient under guardianship or curatorship
* Subjects not covered by public health insurance
* Absence of written informed consent from the patient or his or her proxy (if present) before inclusion or when possible when the patient has been included in an emergency setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-05-23 (Estimated); Study Completion 2026-08-23 (Estimated)

PRIMARY OUTCOMES:
Day-28 mortality | Up to Day-28
  Mortality rates at Day-28

SECONDARY OUTCOMES:
Intubation rate at Day-28 | Day-28
  Proportion of patients requiring invasive mechanical ventilation
Intubation rate at Day-3 | Day-3
  Proportion of patients requiring invasive mechanical ventilation
Intubation rate at Day-7 | Day-7
  Proportion of patients requiring invasive mechanical ventilation
Oxygenation up to Day-7 | Up to Day-7
  Proportion of patients with better oxygenation
Need of other rescue oxygen therapy up to Day-7 | Up to Day-7
  Proportion of patients requiring rescue oxygen therapy
ICU length of stay | Up to Day-90
  Duration time in ICU
Hospital length of stay | Up to Day-90
  Duration time in Hospital
Mortality rates in ICU | Up to Day-90
  Mortality rates in ICU
Mortality rates in hospital | Up to Day-90
  Mortality rates in hospital
Day-90 mortality | Day-90
  Mortality rates at Day-90
Adverse events | Up to Day-90
  Related to the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Samir Jaber, MD, PhD, Study Director — Department of anaesthesia and ICU Saint-Eloi Hospital, Montpellier University Hospital
Locations (1):
- Montpellier University Hospital - Saint Eloi Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
Only the statisticians will have access to the full trial dataset during the enrolment period. All data will be made available to the coordinator at the end of inclusion. Controlled access will be granted to participant-level data sets.
  Technical appendix, statistical code, and dataset will be available on demand.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication, no end date.
Access Criteria: Data will be available for the corresponding author on reasonable request.

REFERENCES:
- [Derived] Jaber S, Huguet H, Molinari N, De Jong A. Comparing high-flow nasal cannula oxygen and non-invasive ventilation to standard oxygenation in non-selected intensive care unit patients admitted for acute hypoxaemic respiratory failure: protocol for the KISS (Key oxygenation Interventions in Surgical and non-Surgical patients) adaptive randomised controlled trial. BMJ Open. 2025 Oct 20;15(10):e100149. doi: 10.1136/bmjopen-2025-100149. PMID 41120174